CLINICAL TRIAL: NCT04289311
Title: SMYLS: A Self-management Program for Youth Living With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shannon Phillips, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00084400
Record Dates: First submitted 2020-02-07; First posted 2020-02-28 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Single group study; all participants are in the intervention arm and receive the intervention
  Interventions: Behavioral: Voice Crisis Alert V2

INTERVENTIONS:
Behavioral: Voice Crisis Alert V2 — An mHealth intervention (app) with multiple components for self-management behavior development. Components include: electronic educational information, symptom monitoring and tracking, communication with a provider, health history entry and storage (including medication adherence).

SUMMARY:
The purpose of this study is to find out whether a web-based intervention using a mobile device is helpful for teens learning to care for and manage symptoms of sickle cell disease. The intervention lasts 12 weeks with a 3-month follow up period, and uses a smartphone or a tablet.

DETAILED DESCRIPTION:
The purpose of the proposed study is to test the feasibility of SMYLS, an mHealth intervention designed to facilitate self-management behaviors in children and adolescents with sickle cell disease (SCD). Specifically, the investigators propose to test the feasibility of the intervention for improving transition from parent-managed to adolescent self-managed care. In addition, the investigators will evaluate the communication that takes place via the intervention between adolescents, their parents/caregivers, and healthcare providers. The investigators will work with the MUSC Pediatric Sickle Cell Clinic to identify and recruit 5 healthcare providers of children with SCD and 30 dyads of adolescents ages 11 - 17 SCD and their parent/caregiver (n = 60).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SCD as reported by provider
* self-reported history of pain at least once per month
* caregiver/parent willingness to participate
* owns a smartphone

Exclusion Criteria:

* not under the care of a provider participant
* cognitive disability or delay that precludes ability to participate, defined as classified severe neurocognitive deficits as documented by neuropsychological evaluation in the medical record
* lack of wi-fi access

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adolescents ages 11 - 17 were enrolled as a dyad with a parent or primary caregiver (n = 30 dyads). 15 young adults ages 18 - 25 were enrolled as individuals. 5 SCD healthcare providers were enrolled.
Groups:
- Intervention Arm: Adolescents 11 - 17 Years; Intervention Arm: Caregivers; Intervention Arm: Young Adults 18 - 25 Years; Healthcare Providers: Single group study; all participants are in the intervention arm and receive the intervention. Arms are designated for adolescents 11 - 17, caregivers of adolescents, young adults 18 - 25, and healthcare providers.
  Voice Crisis Alert V2: An mHealth intervention (app) with multiple components for self-management behavior development. Components include: electronic educational information, symptom monitoring and tracking, communication with a provider, health history entry and storage (including medication adherence).
Period: Overall Study
Arm/Group | Intervention Arm: Adolescents 11 - 17 Years | Intervention Arm: Caregivers | Intervention Arm: Young Adults 18 - 25 Years | Healthcare Providers
Started | 30 | 30 | 15 | 5
Mid-intervention Assessment (6 Weeks) | 25 | 25 | 15 | 5
End-of-intervention Assessment (12 Weeks) | 26 | 26 | 15 | 5
Post-intervention Follow up (24 Weeks) | 24 | 24 | 15 | 5
Completed | 24 | 24 | 15 | 5
Not Completed | 6 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Adolescents 11-17 Years; Intervention Arm: Caregivers; Intervention Arm: Young Adults 18 - 25 Years; Healthcare Providers: Single group study; all participants are in the intervention arm and receive the intervention. Adolescents 11 - 17 years were enrolled as dyads with a parent/primary caregiver (n = 30), young adults were enrolled individually (n = 15), and 5 SCD healthcare providers were enrolled.
  Voice Crisis Alert V2: An mHealth intervention (app) with multiple components for self-management behavior development. Components include: electronic educational information, symptom monitoring and tracking, communication with a provider, health history entry and storage (including medication adherence).
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: Adolescents 11-17 Years | Intervention Arm: Caregivers | Intervention Arm: Young Adults 18 - 25 Years | Healthcare Providers | Total
Number analyzed (Participants) | 30 | 30 | 15 | 5 | 80
Age, Categorical [Count of Participants; unit: Participants] — Population: Healthcare providers were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 30 | 30 | 15 | 0 | 75
    <=18 years | 30 | 0 | 0 |  | 30
    Between 18 and 65 years | 0 | 28 | 15 |  | 43
    >=65 years | 0 | 2 | 0 |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Healthcare providers were not assessed for this baseline measure.
  years
    number analyzed (Participants) | 30 | 30 | 15 | 0 | 75
    (all) | 13.8 (4.7) | 42.6 (10.1) | 20 (2.1) |  | 26 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 30 | 9 | 5 | 58
  Male | 16 | 0 | 6 | 0 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 29 | 30 | 14 | 5 | 78
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 29 | 28 | 15 | 2 | 74
  White | 1 | 1 | 0 | 3 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 15 | 5 | 80
Parent/caregiver type [Count of Participants; unit: Participants] — Population: Healthcare providers, Adolescents, and Young Adults were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 30 | 0 | 0 | 30
    Mother |  | 27 |  |  | 27
    Grandmother |  | 1 |  |  | 1
    missing |  | 2 |  |  | 2
Employment status [Count of Participants; unit: Participants]
  Full-time | 0 | 19 | 1 | 5 | 25
  Part-time | 0 | 4 | 4 | 0 | 8
  Not employed | 0 | 4 | 6 | 0 | 10
  Retired | 0 | 2 | 0 | 0 | 2
  missing | 0 | 1 | 1 | 0 | 2
  Student | 30 | 0 | 3 | 0 | 33
Education level [Count of Participants; unit: Participants] — Population: Healthcare providers were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 30 | 30 | 15 | 0 | 75
    8th grade or less | 16 | 1 | 0 |  | 17
    Some high school | 13 | 2 | 4 |  | 19
    High school graduate | 0 | 6 | 7 |  | 13
    Some college | 0 | 9 | 4 |  | 13
    College graduate | 0 | 7 | 0 |  | 7
    Post graduate or higher level degree | 0 | 4 | 0 |  | 4
    missing | 1 | 1 | 0 |  | 2
Marital status [Count of Participants; unit: Participants] — Population: Healthcare providers were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 30 | 30 | 15 | 0 | 75
    Never married | 30 | 16 | 13 |  | 59
    Married | 0 | 8 | 0 |  | 8
    Widowed | 0 | 1 | 0 |  | 1
    Separated | 0 | 1 | 0 |  | 1
    Divorced | 0 | 2 | 0 |  | 2
    Prefer not to respond | 0 | 1 | 1 |  | 2
    Missing | 0 | 1 | 0 |  | 1
    Resides with SO | 0 | 0 | 1 |  | 1
Household size [Count of Participants; unit: Participants] — Population: Healthcare providers were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 30 | 30 | 15 | 0 | 75
    1 | 1 | 1 | 0 |  | 2
    2 | 2 | 2 | 2 |  | 6
    3 | 8 | 8 | 2 |  | 18
    4 | 7 | 7 | 8 |  | 22
    5 | 8 | 8 | 1 |  | 17
    6 | 1 | 1 | 2 |  | 4
    7 | 1 | 1 | 0 |  | 2
    Prefer not to respond | 1 | 1 | 0 |  | 2
    Missing | 1 | 1 | 0 |  | 2
Type of licensed provider [Count of Participants; unit: Participants] — Population: Adolescents, Caregivers, and Young Adults were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Nurse Practitioner |  |  |  | 2 | 2
    Medical Doctor |  |  |  | 2 | 2
    Physician Assistant |  |  |  | 1 | 1
Primary specialty or subspecialty [Count of Participants; unit: Participants] — Population: Adolescents, Caregivers, and Young Adults were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Hematology |  |  |  | 3 | 3
    Hematology/Oncology |  |  |  | 2 | 2
Years' experience caring for individuals with SCD [Count of Participants; unit: Participants] — Population: Adolescents, Caregivers, and Young Adults were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Less than 10 years |  |  |  | 1 | 1
    10 - 20 years |  |  |  | 1 | 1
    20 or more years |  |  |  | 3 | 3
Number of individual children (<18 years) with SCD seen in the past 12 months [Count of Participants; unit: Participants] — Population: Adolescents, Caregivers, and Young Adults were not assessed for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Less than 200 |  |  |  | 1 | 1
    200 - 300 |  |  |  | 2 | 2
    More than 300 |  |  |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recruitment: Dyads
Description: Number of participant dyads recruited and enrolled per week. (Benchmark is 2 dyads recruited and enrolled per week to reach sample size of 30 dyads)
Time Frame: 6 months
Population: Healthcare providers: Variable not assessed
Measure: Number; unit: dyads recruited and enrolled/week
Groups:
- Adolescent/Caregiver Dyads: Adolescent/caregiver dyads receiving intervention
- Young Adults: Individual young adults receiving intervention
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 30 | 0
dyads recruited and enrolled/week | 2 |

2. Primary Outcome: Participant Adherence to the Intervention
Description: Number of participants (adolescent/caregiver dyads and young adults) using the app from baseline to 6 weeks
Time Frame: baseline to 6 weeks
Population: Healthcare providers did not receive the intervention and are not included in this variable
Measure: Count of Participants; unit: Participants
Groups:
- Adolescents and Caregiver Dyads: Number of dyads receiving intervention
- Young Adults: Number of individual young adults receiving intervention
Arm/Group | Adolescents and Caregiver Dyads | Young Adults
Number analyzed (Participants) | 30 | 15
Participants | 24 | 12

3. Primary Outcome: Consistency of Intervention Delivery
Description: Number of participants (adolescent/caregiver dyads and young adults) to whom instructions on the intervention were provided as recorded in study logs
Time Frame: 24 weeks
Population: Healthcare providers did not receive the intervention and are not included.
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent/Caregiver Dyads: Dyads receiving intervention
- Young Adults: Young adults receiving intervention
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 30 | 15
Participants | 30 | 15

4. Primary Outcome: Projection of Future Adoption
Description: Number of participants (adolescent/caregiver dyads and individual young adults) who report they are likely or very likely to continue using the intervention during post-intervention, semi-structured interviews
Time Frame: 12 weeks
Population: 12 dyads who completed end-of-intervention interview 10 young adults who completed end-of-intervention interview Healthcare providers did not receive the intervention and are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 12 | 10
Participants | 12 | 9

5. Primary Outcome: Participant (Adolescent/Caregiver Dyads and Young Adults) Adherence to the Intervention From 6 Weeks to 12 Weeks
Description: Number of participants (adolescent/caregiver dyads and young adults) who used the intervention from week 6 to week 12
Time Frame: 6 weeks to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Young Adults: Individual young adults receiving the intervention
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 30 | 15
Participants | 16 | 8

6. Primary Outcome: Participant (Adolescent/Caregiver Dyads and Young Adults) Adherence to the Intervention From 12 Weeks to 24 Weeks
Description: Number of participants (adolescent/caregiver dyads and young adults) who used the intervention from week 12 to week 24
Time Frame: 12 weeks to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 30 | 15
Participants | 12 | 4

7. Primary Outcome: Rate of Recruitment: Young Adults
Description: Number of young adult participants recruited and enrolled per week. (Benchmark is 2 young adults recruited per week to reach a sample size of 15).
Time Frame: 6 months
Population: Healthcare providers: variable not assessed
Measure: Number; unit: young adults recruited and enrolled/week
Arm/Group | Adolescent/Caregiver Dyads | Young Adults
Number analyzed (Participants) | 0 | 15
young adults recruited and enrolled/week |  | 4

8. Secondary Outcome: Difference in Mean Pain Score Rating From Baseline to End-of-Intervention
Description: Adolescents: Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference Pediatric Short Form 8a: Change in score at 12 weeks minus baseline. Raw scores range from 0 - 32 with 0 being the lowest pain rating and 32 the highest pain rating. Any decrease in mean difference between scores = improved Young adults: Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference Short Form 8a: Change in score at 12 weeks minus baseline. Raw scores range from 8 - 40 with 8 being the lowest pain rating and 40 the highest pain rating. Any decrease in mean difference between scores = improved
Time Frame: baseline, 12 weeks
Population: Adolescents: 26 participants retained to 12 weeks (end-of-intervention) for analysis Young adults: 15 participants retained to 12 weeks (end-of-intervention) for analysis Caregivers: Variable not assessed Healthcare providers: Variable not assessed
Measure: Mean (95% Confidence Interval); unit: scores on scale
Groups:
- Adolescents: Adolescents receiving intervention
- Young Adults: Young adults receiving the intervention
Arm/Group | Adolescents | Young Adults
Number analyzed (Participants) | 26 | 15
scores on scale | -8.5 [-13.9 to -3.2] | -6.8 [-11.5 to -2.1]

9. Secondary Outcome: Difference in Mean Scores for Transition Readiness From Baseline to End-of-intervention
Description: Adolescents and Young Adults: Assessed using the STARx, in which higher scores indicate greater readiness for transition and the Parent and Youth Sickle Cell Responsibility Scales. Items on the Sickle Cell Responsibility Scales indicate whether parents or children are taking responsibility for health care treatments and are analyzed in conjunction to determine the level of child treatment responsibility, and agreement between the youth and parent for responsibilities. Each item is scored individually and is worth 1 to 5 points. There are 3 subdomains; subdomain scores are summed for the total score, which ranges from 0 - 90 points. Higher scores = improvement
Time Frame: baseline, 12 weeks
Population: Caregivers: variable not assessed Healthcare providers: variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adolescents | Young Adults
Number analyzed (Participants) | 26 | 15
score on a scale | 0.6 [-2.8 to 4.0] | 1.2 [-2.2 to 4.6]

10. Secondary Outcome: Difference in Mean Scores for Anxiety From Baseline to End-of-Intervention
Description: Adolescents: Patient Reported Outcomes Measurement System (PROMIS) Pediatric Short Form Anxiety 8a: Raw Scores range from 0 - 32 with 0 being the lowest anxiety rating and 32 the highest anxiety rating. Change in score at 12 weeks minus baseline. Any decrease difference in mean scores = improved Young adults: Patient Reported Outcomes Measurement System (PROMIS) Short Form Anxiety 8a: Raw Scores range from 8 - 40 with 8 being the lowest anxiety rating and 40 the highest anxiety rating. Change in score at 12 weeks minus baseline. Any decrease difference in mean scores = improved Caregivers: Patient Reported Outcomes Measurement System (PROMIS) Short Form Anxiety 4a: Raw scores range from 4 - 20 with 4 being the lowest anxiety rating and 20 the highest anxiety rating. Change in score at 12 weeks minus baseline. Any decrease difference in mean scores = improved
Time Frame: baseline, 12 weeks
Population: Adolescents and caregivers: 26 dyads retained to 12 weeks and included in the analysis Young adults: 15 participants retained to 12 weeks and included in the analysis Healthcare providers: Variable not assessed
Measure: Mean (95% Confidence Interval); unit: scores on scale
Groups:
- Caregivers: Caregivers participating as a dyad with adolescent
Arm/Group | Adolescents | Young Adults | Caregivers
Number analyzed (Participants) | 26 | 15 | 26
scores on scale | -1.5 [-5.7 to 2.8] | 2.3 [-1.8 to 6.4] | -0.2 [-4.8 to 4.4]

11. Secondary Outcome: Differences in Mean Scores on Depressive Symptoms From Baseline to End-of-Intervention
Description: Adolescents: Patient Reported Outcomes Measurement System (PROMIS) Pediatric short form depression 8a: Raw scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Change in score at 12 weeks minus baseline. Any decrease in differences in mean scores = improved Young Adults: Patient Reported Outcomes Measurement System (PROMIS) short form depression 8a: Raw scores range from 8 - 40, with 8 being the lowest depression rating and 40 the highest depression rating. Change in score at 12 weeks minus baseline. Any decrease in differences in mean scores = improved Caregivers: Patient Reported Outcomes Measurement System (PROMIS) depression 4a: Raw scores range from 4 - 20, with 4 being the lowest depression rating and 20 the highest depression rating. Change in score at 12 weeks minus baseline. Any decrease in differences in mean scores = improved
Time Frame: baseline, 12 weeks
Population: Healthcare providers: Variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Caregivers: Caregivers participating with adolescent as a dyad
Arm/Group | Adolescents | Young Adults | Caregivers
Number analyzed (Participants) | 26 | 15 | 26
score on a scale | -1.4 [-5.4 to 2.6] | -2.2 [-7.5 to 3.1] | 0.8 [-2.1 to 3.8]

12. Secondary Outcome: Differences in Mean Scores for Pain Intensity From Baseline to End-of-interention
Description: Adolescents: Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity Pediatric 3a. Raw scores range from 3 - 15, with 3 being the lowest pain intensity rating and 15 being the highest pain intensity rating. Change in score at 12 weeks minus baseline. Any decrease in mean difference between scores = improved.
  Young adults: Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity v2 3a. Raw scores range from 3 - 15, with 3 being the lowest pain intensity rating and 15 being the highest pain intensity rating. Change in score at 12 weeks minus baseline. Any decrease in mean difference between scores = improved.
Time Frame: baseline, 12 weeks
Population: Caregivers: Variable not assessed Healthcare providers: Variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adolescents | Young Adults
Number analyzed (Participants) | 26 | 15
score on a scale | -2.7 [-7.1 to 1.8] | -3.8 [-9.0 to 1.5]

13. Secondary Outcome: Difference in Mean Scores for Fatigue From Baseline to End-of-Intervention
Description: Adolescents: Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Pediatric Short Form 10a: Raw scores range from 0 - 40 with 0 being the least amount of fatigue and 40 the most fatigue. Difference in mean scores at 12 weeks minus baseline. Any decrease in rating = improved Young Adults: Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a: Raw scores range from 8 - 40 with 8 being the least amount of fatigue and 40 the most fatigue. Difference in mean scores at 12 weeks minus baseline. Any decrease in rating = improved Caregivers: Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 4a: Raw scores range from 4 - 20 with 4 being the least amount of fatigue and 20 the most fatigue. Difference in mean scores at 12 weeks minus baseline. Any decrease in rating = improved
Time Frame: baseline, 12 weeks
Population: Healthcare providers: Variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Caregivers: Caregivers participating with adolescents as dyad
Arm/Group | Adolescents | Young Adults | Caregivers
Number analyzed (Participants) | 26 | 15 | 26
score on a scale | -0.7 [-3.8 to 2.5] | -5.2 [-9.8 to -0.6] | 2.3 [-1.1 to 5.8]

14. Secondary Outcome: Differences in Mean Scores for Quality of Life From Baseline to End-of-Intervention
Description: Adolescents: Pediatric Quality of Life Inventory (Peds QL): Scores are transformed on a scale from 0 - 100, with 0 indicating the highest possible problems with quality of life and 100 indicating the lowest possible problems with quality of life. Change in score at 12 weeks minus baseline. Any increase in difference between mean scores = improved.
  Caregivers: Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Physical: Raw scores range from 4 - 20 with 4 being the lowest global physical health and 20 the highest global physical health. Difference in mean scores at 12 weeks minus baseline. Any increase in rating = improved
Time Frame: baseline, 12 weeks
Population: Young Adults: Only condition-specific health-related quality of life was assessed and is reported in outcome number 14.
  Healthcare providers: variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adolescents | Caregivers
Number analyzed (Participants) | 26 | 26
score on a scale | 0.9 [-4.1 to 6.0] | -3.4 [-6.2 to -0.6]

15. Secondary Outcome: Differences in Mean Scores for Condition-Specific Quality of Life From Baseline to End-of-Intervention
Description: Adolescents: Pediatric Quality of Life Inventory (PedsQL) with SCD module: Scores are transformed on a scale from 0 - 100, with 0 indicating the highest possible problems with quality of life and 100 indicating the lowest possible problems with quality of life. Change in score at 12 weeks minus baseline. Any increase in difference in means scores = improved.
  Young Adults: Adult Sickle Cell Disease Quality of Life Information System (ASCQ-Me): Raw scores for each scale (emotional impact, social impact, sleep impact, stiffness impact, pain impact) range from 5 to 25 with 5 being the lowest health-related quality of life score for each and 25 the highest. Change in score at 12 weeks minus baseline. Any increase in difference in means scores = improved.
Time Frame: baseline, 12 weeks
Population: Caregivers: variable not assessed Healthcare providers: variable not assessed Young adults were not assessed with the PedsQL SCDM and adolescents were not assessed with the ASCQ-Me.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adolescents | Young Adults
Number analyzed (Participants) | 26 | 15
score on a scale
  PedsQL SCDM Total score: number analyzed (Participants) | 26 | 0
  PedsQL SCDM Total score | 7.2 [2.6 to 11.9] |
  ASCQ-Me Emotional Impact: number analyzed (Participants) | 0 | 15
  ASCQ-Me Emotional Impact |  | 2.2 [0.0 to 4.3]
  ASCQ-Me Social Impact: number analyzed (Participants) | 0 | 15
  ASCQ-Me Social Impact |  | 7.4 [2.3 to 12.4]
  ASCQ-Me Sleep Impact: number analyzed (Participants) | 0 | 15
  ASCQ-Me Sleep Impact |  | 2.7 [-1.0 to 6.4]
  ASCQ-Me Stiffness Impact: number analyzed (Participants) | 0 | 15
  ASCQ-Me Stiffness Impact |  | 3.1 [-1.9 to 8.0]
  ASCQ-Me Pain Impact: number analyzed (Participants) | 0 | 15
  ASCQ-Me Pain Impact |  | 6.1 [1.7 to 10.5]

16. Secondary Outcome: Difference in Mean Scores for Self-Efficacy From Baseline to End-of-Intervention
Description: Adolescents and Young Adults: Sickle Cell Self-Efficacy Scale: Raw scores range from 9 to 45, with 9 being the lowest self-efficacy rating and 45 the highest. Change in score at 12 weeks minus baseline. Any increase in scores = improved
Time Frame: baseline, 12 weeks
Population: Caregivers: variable not assessed Healthcare providers: variable not assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adolescents | Young Adults
Number analyzed (Participants) | 26 | 15
score on a scale | -0.6 [-4.4 to 3.1] | 0.4 [-4.2 to 5.0]

ADVERSE EVENTS:
Time Frame: Duration of study participation: 24 weeks
Groups:
- Adolescents: Adolescents ages 11 - 17 years receiving intervention
- Caregivers: Caregivers of adolescents participating as a dyad
- Young Adults: Young adults ages 18 - 25 receiving intervention
- Healthcare Providers: Healthcare providers participating in study
Arm/Group | Adolescents | Caregivers | Young Adults | Healthcare Providers
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/30 | 0/30 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/15 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (N=30) | Caregivers (N=30) | Young Adults (N=15) | Healthcare Providers (N=5)
Hospitalization for vasoocclusive episode (Blood and lymphatic system disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (N=30) | Caregivers (N=30) | Young Adults (N=15) | Healthcare Providers (N=5)
Vasoocclusive episode without hospitalization (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of this feasibility study included measurement issues with the clinic appointment attendance. We were unable to assess this outcome measure with accuracy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT04289311/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT04289311/ICF_001.pdf